CLINICAL TRIAL: NCT05283811
Title: Mapping Algorithmic State Space in the Human Brain
Brief Title: Understanding Prefrontal and Medial Temporal Neuronal Responses to Algorithmic Cognitive Variables in Epilepsy Patients
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Baylor College of Medicine (Other)
Responsible Party: Principal Investigator, Sameer Sheth, Associate Professor, Baylor College of Medicine
Allocation: Non-Randomized | Model: Factorial | Masking: None | Purpose: Health Services Research
Other Study IDs: H18112
Record Dates: First submitted 2022-02-28; First posted 2022-03-17 (Actual); Last update posted 2025-07-20 (Actual); Status verified 2025-07

CONDITIONS: Epilepsy
Keywords: Single-neuron; Local-field potentials
MeSH Terms: conditions — Epilepsy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Epilepsy Monitoring Unit (Other): Patient's behavioral and neural activity via computer tasks and questionnaires are monitored in the Epilepsy Monitoring Unit
  Interventions: Behavioral: EMU
- Neuropace RNS Device (Other): Patients are implanted with RNS device to treat their seizure activity
  Interventions: Device: NEUROPACE RNS SYSTEM

INTERVENTIONS:
Device: NEUROPACE RNS SYSTEM — This device is indicated as a therapy in reducing the frequency of seizures in individuals
  Arms: Neuropace RNS Device
Behavioral: EMU — Patients are admitted to the Epilepsy Monitoring Unit for observation of seizure activity prior to further treatment
  Arms: Epilepsy Monitoring Unit

SUMMARY:
Humans have a remarkable ability to flexibly interact with the environment. A compelling demonstration of this cognitive flexibility is human's ability to respond correctly to novel contextual situations on the first attempt, without prior rehearsal. The investigators refer to this ability as 'ad hoc self-programming': 'ad hoc' because these new behavioral repertoires are cobbled together on the fly, based on immediate demand, and then discarded when no longer necessary; 'self-programming' because the brain has to configure itself appropriately based on task demands and some combination of prior experience and/or instruction. The overall goal of our research effort is to understand the neurophysiological and computational basis for ad hoc self-programmed behavior. The previous U01 project (NS 108923) focused on how these programs of action are initially created. The results thus far have revealed tantalizing notions of how the brain represents these programs and navigates through the programs. In this proposal, therefore, the investigators focus on the question of how these mental programs are executed. Based on the preliminary findings and critical conceptual work, the investigators propose that the medial temporal lobe (MTL) and ventral prefrontal cortex (vPFC) creates representations of the critical elements of these mental programs, including concepts such as 'rules' and 'locations', to allow for effective navigation through the algorithm. These data suggest the existence of an 'algorithmic state space' represented in medial temporal and prefrontal regions. This proposal aims to understand the neurophysiological underpinnings of this algorithmic state space in humans. By studying humans, the investigators will profit from our species' powerful capacity for generalization to understand how such state spaces are constructed. The investigators therefore leverage the unique opportunities available in human neuroscience research to record from single cells and population-level signals, as well as to use intracranial stimulation for causal testing, to address this challenging problem. In Aim 1 the investigators study the basic representations of algorithmic state space using a novel behavioral task that requires the immediate formation of unique plans of action. Aim 2 directly compares representations of algorithmic state space to that of physical space by juxtaposing balanced versions of spatial and algorithmic tasks in a virtual reality (VR) environment. Finally, in Aim 3, the investigators test hypotheses regarding interactions between vPFC and MTL using intracranial stimulation.

ELIGIBILITY:
Inclusion Criteria:

* Eligible subjects include both male and female patients, between 10 years of age and 64 years of age, who undergo placement of intracranial electrodes for clinical characterization of epilepsy.

Exclusion Criteria:

* Grounds for exclusion would include inability to understand and follow instructions, or inability to concentrate sufficiently to achieve a high proportion of correct responses.

Ages: 10 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 205 (Estimated)
Dates: Start 2021-06-01 (Actual); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
Behavioral performance (Accuracy as fraction of correct responses) | 7-14 days of behavioral performance collection
  Patients will be asked to perform a few different novel, computerized tasks where the patients must respond to on-screen stimuli using button presses. Behavior will be assessed in terms of the accuracy of these responses.
Neurophysiological activity (single-neuron activity in spikes/second) | 7-14 days of neural activity collection
  While patients are performing each behavioral task, the investigators will measure neural activity from BlackRock using depth electrodes with the aim of isolating single-neuron activity (for patients in the EMU) and local-field potential activity (for patients in the RNS patients). Neurophysiological activity will be analyzed with the aim of understanding the neural representations underlying cognitive performance during the task.

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - University of California, Los Angeles, Los Angeles, California
  - Baylor College of Medicine, Houston, Texas
  - University of Utah, Salt Lake City, Utah